CLINICAL TRIAL: NCT00097682
Title: Ethics Study to Understand the Views of Cancer Patients Regarding Financial Conflicts of Interest in Research
Brief Title: Views of Cancer Patients Regarding Financial Conflicts of Interest
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050038; 05-CC-0038
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-02

CONDITIONS: Neoplasms
Keywords: Financial Ties; Institution; Research Doctor; Oncology; Attitudes; Cancer; Survey
MeSH Terms: conditions — Neoplasms; Behavior

SUMMARY:
This study will explore what research patients understand about financial collaborations in the research setting and their concerns about these collaborations. Financial partnerships are crucial to advancing medical research; however, they are giving rise to increasing concerns about financial conflicts of interest and possible impacts on the integrity of research and patient safety. This study will examine patients' views about financial ties between drug companies and the doctors running research studies, as well as ties between the drug companies and the cancer centers where the studies are conducted.

Patients 18 years of age and older who are enrolled in cancer studies at the National Cancer Institute in Bethesda, MD; the Fred Hutchinson Cancer Research Center in Seattle, WA; the Dana-Farber Cancer Institute in Boston, MA; the Columbia Comprehensive University Herbert Irving Cancer Center in New York, NY; and the University of Colorado Cancer Center in Denver, CO, may be eligible for this study.

Participants are interviewed about the following:

* Patients' awareness and understanding about individual and institutional financial conflicts of interest, and how such conflicts, if they exist, are being managed
* The impact of a researcher's financial ties on the patient's decision to participate in that researcher's study
* The impact of the institution's financial ties on the patient's decision to participate in research at that institution
* Attitudes about policies and practices regarding conflicts of interest in the research setting
* Attitudes about disclosure of conflicts of interest in the research setting
* Patient symptoms and performance
* Patient's cancer trial
* Patient's cancer history
* Patient's trust
* Patient demographics (gender, age, race, religion, education, income, health insurance, employment).

DETAILED DESCRIPTION:
This study seeks to inform deliberation of ethical issues related to financial conflicts of interest in clinical research through empirical data obtained from patients participating in cancer studies. In particular, this study endeavors to describe and summarize the views of patients about both individual and institutional financial conflicts of interest pertaining to clinical research. This study will assess awareness of financial conflicts of interest and the current safeguards in place to manage financial ties; assess the impact of hypothetical financial conflicts of interest on a research subject's decision to participate in a clinical study; identify the reasons that financial conflicts of interest either do or do not influence patients' research participation; summarize views regarding the presence of financial conflicts of interest and what limits should be in place to manage them; identify interests about disclosure of these financial conflicts of interest; describe demographic characteristics of subjects enrolled in the survey and evaluate the impact of demographic information on subjects' views regarding financial conflicts of interest. Participants will be recruited from all phases of oncology studies being conducted at 5 sites, the National Cancer Institute in Bethesda, MD; the Dana-Farber Cancer Institute in Boston, MA; the Fred Hutchinson Cancer Research Center in Seattle, WA; the University of Colorado Cancer Center in Denver, CO, and the Columbia University Herbert Irving Comprehensive Cancer Center in New York, NY. The primary methodology for the study is an in-person administration of a questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be included if they:

1. Have consented to participate in a phase I, I/II, II, or III cancer study and are at any point in that study.
2. Give informed consent.
3. Understand written and spoken English.
4. Are over 18 years of age.

EXCLUSION CRITERIA:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-11-18; Study Completion 2007-10-02

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Kelch RP. Maintaining the public trust in clinical research. N Engl J Med. 2002 Jan 24;346(4):285-7. doi: 10.1056/NEJM200201243460413. No abstract available. PMID 11807156